CLINICAL TRIAL: NCT05760404
Title: Modulatory Effects of Active Drugs on the Endocannabinoid System on Spontaneous and Induced Contractility of the Colon
Acronym: CB1 - CONTRACT
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PERSIANI ROBERTO, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5309
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgery for colorectal cancer — Patients undergoing upfront surgery or surgery after neoadjuvant therapy for colorectal cancer with curative intention
Other: in vitro study — on tissues from colorectal resections

SUMMARY:
The endocannabinoid system plays important roles in the modulation of gastrointestinal motility and secretions. These effects are mainly mediated by the activation by the endocannabinoids anandamide (AEA) and 2-arachidonylglycerol (2-AG) of CB1 receptors expressed on cholinergic neurons. Cannabis sativa extracts also perform these activities, through the detection of CB1 receptors by the phytocannabinoids they contain, in particular delta9-tetrahydrocannabinol.

CB1 receptors are abundantly expressed at the synaptic terminals of excitatory motor neurons and cholinergic secretomotor neurons and their activation induces prejunctional inhibition of acetylcholine release. It is thought that the endocannabinoids AEA and 2-AG, by activating these receptors, may exert a physiological control on gastrointestinal contractility and secretions.

This research hypothesizes that drugs capable of inhibiting the biosynthetic and catabolic enzymes of endocannabinoids, of inhibiting the transmembrane transport of endocannabinoids or of allosterically modulating CB1 receptors induce important regulating effects of basal contractility and excitatory motor responses, induced by activation of neurons intramural cholinergics, of colonic circular smooth muscle.

The effects of drugs acting on CB receptors, endocannabinoid biosynthetic and catabolic enzymes and endocannabinoid membrane transporters on basal contractility or induced by neuronal activation of colonic preparations in vitro will be evaluated.

The study will enroll patients affected by colorectal cancer to undergo elective resective surgery at any stage, undergoing upfront surgery or after neo-adjuvant therapy with a therapeutic interval greater than 6 weeks. In the selected patients (see inclusion/exclusion criteria), a fresh sample of about 2.5 cm of healthy colon (healthy resection margin) will be taken, which will be taken in the operating room and sent to the laboratory for in vitro study.

Expected results: The study is expected to provide new evidence regarding the induction of pharmacological effects by allosteric receptor modulators of CB1 receptors, inhibitors of endocannabinoid biosynthetic and catabolic enzymes, and inhibitors of cannabinoid transporters in the human colon, which may open interesting perspectives regarding the development of new therapeutic strategies for the treatment of constipation, diarrhea and irritable bowel syndrome.

DETAILED DESCRIPTION:
The present research is aimed at defining the roles of the different components of the endocannabinoid system in the regulation of the basal contractile activity and of the excitatory motor responses induced by neuronal activation in the human colon.

Therefore, the motor effects of drugs acting on the various components of this system will be evaluated, ie receptors, biosynthetic and catabolic enzymes and membrane transporters, in colonic preparations, in conditions of basal muscle tone and on muscle contractions induced by neuronal activation.

If the modulation of one or more components of the endocannabinoid system proves to be important in the regulation of colonic contractility and probably useful for therapeutic purposes, drugs active on them could represent new treatments for constipation, diarrhea or some forms of irritable bowel syndrome, very common in the gastrointestinal tract.

Particular interest will be focused on the effects of allosteric modulators of CB1 receptors, inhibitors of biosynthetic and catabolic enzymes of endocannabinoids and inhibitors of membrane transporters of endocannabinoids.

This is an exploratory study, in which pre-specified hypotheses on pre-specified sample sizes will not be tested. Therefore, the data will be subjected only to descriptive statistics, without conducting any tests of statistical significance on them. Consequently, no primary or secondary endpoints are foreseen.

ELIGIBILITY:
Inclusion Criteria:

* patients with colorectal cancer at any stage of the disease, undergoing upfront surgery or neo-adjuvant therapy for more than 6 weeks, to undergo surgery with resective intent at the UOC of General Surgery 1 of the Fondazione Policlinico Universitario A. Gemelli of Rome in the two years following the approval of the study by the Ethics Committee;

Exclusion Criteria:

* patients with diverticular stenosis, patients with stenosing colorectal cancer (defined as a tumor that cannot be passed through endoscopically, resulting in clinical and/or radiological symptoms of intestinal obstruction), urgent/emergency procedures, patients treated with corticosteroid therapy for immuno-rheumatic diseases, patients treated with radio-chemotherapy and undergone surgery for less than 6 weeks, surgically resected patients who present macroscopic lesions near the resection margin when opening the surgical piece, refusal of informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colorectal cancer at any stage of the disease
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the motor effects of drugs that act on the various components of this system | 30 months
  Evaluate the motor effects of drugs that act on the various components of this system, like receptors, biosynthetic and catabolic enzymes and membrane transporters, in colic tissues, in conditions of basal muscle tone and on muscle contractions induced by neuronal activation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided